CLINICAL TRIAL: NCT02944279
Title: Neutrophil Elastase and Elafin as Prognostic Biomarker for Acute Respiratory Distress Syndrome
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Beijing Friendship Hospital (Other); Beijing Shijitan Hospital, Capital Medical University (Other); Beijing Xiyuan Hospital (Unknown); China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Xi Zhu, Professor, Peking University Third Hospital
Other Study IDs: 2009-1014
Record Dates: First submitted 2016-10-21; First posted 2016-10-25 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Acute Respiratory Distress Syndrome, ARDS
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (5):
- Peking University Third Hospital
- Beijing Friendship Hospital
- Beijing Shijitan Hospital
- Beijing Xiyuan Hospital
- China-Japan Friendship Hospital

SUMMARY:
The acute respiratory distress syndrome (ARDS), characterized by alveolar flooding with protein-rich pulmonary edema fluid, is one of the most common disease in the intensive care unit (ICU) throughout the world. In recent years, much effort has been focused on the biological markers for their potential values to diagnose ARDS and outcomes.

ARDS is generally accompanied by the disruption in alveolar-capillary barrier permeability, which subsequently caused an influx of neutrophils into the interstitium and alveolar space. It was reported that the aggregation, adhesion activation and release proteases of neutrophils are the key pathogenesis of ARDS pulmonary edema. Neutrophil Elastase (HNE), the most crucial protease generated in neutrophil azurophilic granules, plays an important role in various inflammations, especially the lung injury. The destructive action of HNE on almost all extracellular matrix influences cell signaling through cleavage of surface receptors. Once released in circulation, HNE is rapidly inactivated by conjugation with PI3. This local inhibitor reduces HNE mediated tissue injury and inflammation. Thus, the investigators plan to conduct a cohort study with repeated measures to examine the diagnostic and prognostic value of HNE and PI3 for ARDS.

ELIGIBILITY:
Exclusion Criteria:

* Age <18 years
* History of chronic lung diseases, such as interstitial pulmonary fibrosis or bronchiolitis
* history of pneumonectomy
* Treatment with immunomodulating therapy other than corticosteroids, such as granulocyte colony stimulating factor, cyclophosphamide, cyclosporine, interferon, or TNF-α antagonists
* Presence of other immunodeficient conditions, such as HIV infection, leukemia, or neutropenia (absolute neutrophil count <1000/μl)
* History of organs or bone marrow transplant other than autologous bone marrow transplant
* Directive to withhold intubation
* ICU stay duration<72h
* Patient developed ARDS before ICU admission. Sepsis and septic shock were defined according to the Berlin definition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is from five clinical and surgical ICUs in Beijing metropolitan area: Peking University Third Hospital in the northwest of Beijing, Beijing Friendship Hospital in the south, Beijing Shijitan Hospital in the middle, Beijing Xiyuan Hospital in the west, and China-Japan Friendship Hospital in the northeast.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2011-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
ARDS development-Berlin definition | 60 days
ARDS survival | 60 days

IPD SHARING:
Plan to Share IPD: No